CLINICAL TRIAL: NCT00493194
Title: Interstitial Fibrosis in Protocol Biopsies of Renal Allografts: A Prospective, Randomised Trial of Sirolimus Versus Cyclosporine.(Fibrasic)
Brief Title: Fibrosis in Renal Allografts
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-004115-38
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2005-10

CONDITIONS: Kidney Failure, Chronic; Transplantation; Immunosuppression; Interstitial Fibrosis
Keywords: Cyclosporine toxicity; Interstitial Fibrosis; Chronic allograft nephropathy; Sirolimus
MeSH Terms: conditions — Kidney Failure, Chronic; Pulmonary Fibrosis | interventions — Sirolimus; Cyclosporine; Daclizumab

INTERVENTIONS:
Drug: sirolimus
Drug: cyclosporine
Drug: daclizumab

SUMMARY:
This prospective, randomized study, comparing sirolimus to cyclosporine in renal transplant recipients, has two major objectives:

1. -To determine the incidence and the degree of interstitialfibrosis and arteriosclerosis, as wel as the glomerular volume in protocol biopsies at 6 months in sirolimus-and in cyclosporine-treated renal allograft recipients, by means of quantitative computerized image analysis.

   * To determine the prognostic implication of these morphologic changes.
2. To study the expression of genes, involved in inflammation and fibrosis, in protocol biopsies at 6 months in sirolimus-and cyclosporine-treated renal allograft recipients.

DETAILED DESCRIPTION:
Calcineurin inhibitors have significantly improved the one-year graft survival of renal allografts. However, chronic nephrotoxicity caused by calcineurin inhibitors contributes to the long-term decline in renal function in kidney transplant recipients. Approximately ninety percent of the protocol biopsies of renal allografts, performed at 18 months post transplantation, show histological lesions of chronic calcineurin nephrotoxicity . In recent years, two new non-nephrotoxic immunosuppressive drugs, i.e. mycophenolate mofetil and sirolimus, have become available for the prophylaxis of graft rejection in renal transplantation.

Three randomized clinical trials, comparing cyclosporine with sirolimus in combination with mycophenolate mofetil, reported a superior graft function at one year in sirolimus treated renal allograft recipients. However, data on long-term graft survival and histological lesions of protocol biopsies in sirolimus-treated renal transplant recipients, are currently lacking.

In analogy with previous observations in native kidney disease, Grimm et al. recently reported that interstitial fibrosis in protocol biopsies of renal allografts, at 6 months post transplantation, significantly inversely correlates with the subsequent graft survival One hundred recipients of a first renal allograft will be randomized to an immunosuppressive protocol based on cyclosporine (50 patients) or sirolimus (50 patients). Concommittant immunosuppression will be similar in both groups, and consists of Daclizumab as induction treatment (five iv gifts every two weeks), and mycophenolate mophetil and steroids as maintenance immunosuppression.

Randomization will be performed by centre to avoid centre-related bias. All patients will complete a follow-up of 12 months. Two core biopsies of the graft will be obtained in each recipient, at implantation and at 6 months. Serum creatinine and the estimated creatinine clearance (by the Nankivell and the Jellife method) will be monthly recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Recipients of a renal allograft, with a minimum age of 18 years.
2. Male or female recipients. Women of child-bearing age must practice adequate contraception
3. For renal allografts from living donors, at least one HLA-mismatch is required.
4. Written informed consent, compliant with local regulations.

Exclusion Criteria:

1. Recipients of a second or third renal allograft, with a past history of graft failure due to rejection.
2. Recipients of a renal allograft from a haplotype-identical living donor or a non-heart beating donor.
3. Cold ischemia time > 24 hours
4. Recipients of a kidney from donors ≥ 65 years of age
5. Recipients of multiple organs.
6. Pregnant women.
7. Immunological high-risk recipients, defined as current or historical PRA > 50 %
8. Recipients with focal segmental sclerosis as primary renal disease.
9. Recipients with leucopenia (WBC < 3000/mmÂ³), thrombocytopenia (Thr < 100.000/mmÂ³),or hyperlipidemia (Tot Chol > 300 mg/dl or Triglycerides > 300 mg/dl)
10. Previous history of malignancy, except completely excised basocellular skin tumor
11. Chronic active infection.
12. Inadequate compliance to treatment.
13. Use of specific drugs: Terfenadine, pimozide, astemizole, fluconazole, ketoconazole and cimetidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-05; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
The primary end-point of this study will be the cortical fractional interstitial fibrosis volume (V IntFib) in protocol biopsies at 6 months. The V IntFib will be determined on Sirius red stained slides by means of a computerized image analysis program,

SECONDARY OUTCOMES:
Secundary end-points:
-Patient and graft-survival at one year.
-The serum creatinine and the estimated creatinine
clearance at 6 and 12 months.
-The 24 hour proteinuria at 6 and 12 months.
-The intimal area and arterial wall thickness in protocol
biopsies at 6 months.
-The glomerular volume in protocol biopsies at 6 months.
-The incidence of acute rejection episodes during the
first year.
-The severity of acute rejection episodes according to
the Banffâ 97 classification.
-The incidence of infectious complications.
-The incidence of hematological adverse effects.
-The number of antihypertensive and lipid-lowering drugs
at 6 and 12 months.
-The incidence of treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Bosmans, M.D. Ph.D., Principal Investigator — University Hospital, Antwerp
Locations (3):
- Belgium (3):
  - University Hospital Antwerp, Edegem, Antwerp
  - University Hospital Brussels, Brussels (Jette), Brabant
  - University Hospital Gent, Ghent, Oost-Vlaanderen

REFERENCES:
- [Result] Flechner SM, Goldfarb D, Modlin C, Feng J, Krishnamurthi V, Mastroianni B, Savas K, Cook DJ, Novick AC. Kidney transplantation without calcineurin inhibitor drugs: a prospective, randomized trial of sirolimus versus cyclosporine. Transplantation. 2002 Oct 27;74(8):1070-6. doi: 10.1097/00007890-200210270-00002. PMID 12438948
- [Result] Groth CG, Backman L, Morales JM, Calne R, Kreis H, Lang P, Touraine JL, Claesson K, Campistol JM, Durand D, Wramner L, Brattstrom C, Charpentier B. Sirolimus (rapamycin)-based therapy in human renal transplantation: similar efficacy and different toxicity compared with cyclosporine. Sirolimus European Renal Transplant Study Group. Transplantation. 1999 Apr 15;67(7):1036-42. doi: 10.1097/00007890-199904150-00017. PMID 10221490
- [Result] Kreis H, Cisterne JM, Land W, Wramner L, Squifflet JP, Abramowicz D, Campistol JM, Morales JM, Grinyo JM, Mourad G, Berthoux FC, Brattstrom C, Lebranchu Y, Vialtel P. Sirolimus in association with mycophenolate mofetil induction for the prevention of acute graft rejection in renal allograft recipients. Transplantation. 2000 Apr 15;69(7):1252-60. doi: 10.1097/00007890-200004150-00009. PMID 10798738
- [Result] Grimm PC, Nickerson P, Gough J, McKenna R, Stern E, Jeffery J, Rush DN. Computerized image analysis of Sirius Red-stained renal allograft biopsies as a surrogate marker to predict long-term allograft function. J Am Soc Nephrol. 2003 Jun;14(6):1662-8. doi: 10.1097/01.asn.0000066143.02832.5e. PMID 12761269